CLINICAL TRIAL: NCT05028777
Title: Cohort of Patients With Left Ventricular Thrombus: Management and Outcomes in the Direct Oral Anticoagulants Era
Acronym: LV-Thrombus
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-02187
Record Dates: First submitted 2021-08-25; First posted 2021-08-31 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Thrombus of Left Ventricle
Keywords: Left Ventricular Assist Device; Acute Myocardial Infarction; Left Ventricular or Left Ventricle; Dual Antiplatelet Therapy; Direct Oral Anticoagulant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients diagnosed with left ventricular thrombus: All patients diagnosed with left ventricular thrombus through different imaging modalities (echocardiography, CT or MRI) and who have been diagnosed and/or treated at the Inselspital or another site of the Insel Gruppe.

SUMMARY:
The investigators' primary objective is to assess whether a difference in the occurrence of bleeding events exist between patients with LVT treated with DOACs as compared to those treated with VKAs.

DETAILED DESCRIPTION:
Left ventricular thrombus (LVT) is a well-known complication of left ventricle (LV) systolic dysfunction that can be seen in acute systolic dysfunction, i.e. induced by an acute myocardial infarction (AMI) or Takotsubo cardiomyopathy, and in chronic heart failure with reduced ejection fraction (HFrEF), whatever the cause.

Improvements in the management of AMI, particularly with the implementation of primary percutaneous coronary intervention (PCI), have led to a striking reduction in the occurrence of LVT in patients with AMI from about 30% in the thrombolytic era to about 4% nowadays, according to echocardiographic assessment. On the other hand prognosis of patients with LVT didn't change over time: mortality and risk of embolic events associated with this condition are still high.

A limited amount of evidence shows that oral anticoagulation is associated in the majority of patients with both resolution of LVT and reduction in ischemic events. This benefit comes at the cost of bleeding complications, which have been demonstrated to impact on mortality, especially in patients after AMI receiving an oral anticoagulant on top of a dual antiplatelet therapy (so-called triple antithrombotic therapy).

Current European and American guidelines on treatment of myocardial infarction with ST-elevation do not make strong recommendations for the management of LVT, whereas guidelines on treatment of heart failure do not give any. The European Society of Cardiology recommends an anticoagulation treatment for up to 6 months from diagnosis in case of LVT thrombus after AMI and the decision to continue the therapy after 6 months should be taken on the basis of echocardiographic follow-up (class IIa level of evidence C). The American College of Cardiology and American Heart Association (AHA) gives a similar recommendation (IIaC), however specifically mentioning vitamin K antagonists (VKAs) and a target INR (international normalized ratio) 2.0-2.5 for 3 months on top of dual antiplatelet therapy (DAPT). They also propose to consider an anticoagulant therapy for patients with severe anterior wall motion after STEMI but without LVT (IIbC). The AHA and American Stroke Association published in 2014 their last recommendations for secondary stroke prevention, which are in line with the above mentioned guidelines. Direct oral anticoagulants (DOACs) are mentioned as an alternative to VKAs (IIbC).

All guidelines agree that DOACs for LVT treatment cannot be recommended as first-line therapy because of the scarce evidence, based on case reports small case series and only one large retrospective study (RED VELVT study, published on April 22, 2020).

However, in clinical practice because of the establishment of DOACs over VKAs as first-line therapy to prevent embolic events in patients with atrial fibrillation, those are prescribed off-label to a significant number of patients with LVT. DOACs, as compared to VKAs, showed a greater efficacy regarding prevention of ischemic and hemorrhagic stroke and systemic embolic events in atrial fibrillation, but an increased risk of gastrointestinal bleedings.

The pathophysiology of thrombus formation in a left ventricle with regional wall motion abnormalities and in left atrium with atrial fibrillation is very similar and it implies a blood stasis as main mechanism. Thus one could expect that DOACs, which have been demonstrated to be superior to VKAs in term of prevention of embolic events in atrial fibrillation, have a similar effect on treatment of LVT. However, the first large retrospective study including 541 patients with LVT, of which 421 treated with anticoagulation showed an increased risk of embolic events at 1 year among patients with LVT treated with DOACs as compared to those on VKAs; occurrence of bleeding events was not reported.

Beside the above mentioned uncertainty concerning duration and type of treatment (VKAs versus DOACs) in LVT, there are also some issues concerning the imaging modality used for the diagnosis of LVT. Several studies comparing the diagnostic performance of transthoracic echocardiography (TTE) versus cardiac magnetic resonance (CMR) showed a roughly 30% sensitivity of TTE when taking delayed-enhancement CMR (DE-CMR) as gold standard. With the growing use of CMR, an increasing number of patients are diagnosed with small left ventricular thrombi, which would have been missed in usual clinical practice and which seem to be associated with an embolic risk similar to thrombi detected by TTE.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years old at enrolment
* With a LVT identified at echocardiography, MRI or CT between January 1st, 2013 and July 31st, 2020
* Treated at least once at the Inselspital or in another site of the Insel Gruppe
* Able to provide a written informed consent

Exclusion Criteria:

* Documented refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is an observational, retrospective and prospective, monocentric study including all patients diagnosed with left ventricular thrombus through different imaging modalities (echocardiography, CT or MRI)
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
The occurrence at 1 year of bleeding | 1 year
  Primary combined endpoint includes the occurrence at 1 year of bleeding BARC (Bleeding Academic Research) Consortium type 2, 3 or 5.

SECONDARY OUTCOMES:
Rate of patients with arterial systemic embolic event | 1, 2 and 5 years
  Combined endpoint of arterial systemic embolic event, including ischemic stroke, myocardial infarction, peripheral embolism (e.g. splenic infarction, renal infarction, bowel infarction, acute embolic limb ischemia) at 1, 2 and 5 years.
Rate of patients with ischemic stroke | 1, 2 and 5 years
  Each arterial systemic embolic event considered separately at 1, 2 and 5 years
Rate of patients with myocardial infraction | 1, 2 and 5 years
  Each arterial systemic embolic event considered separately at 1, 2 and 5 years
Rate of patients with peripheral embolism | 1, 2 and 5 years
  Each arterial systemic embolic event considered separately at 1, 2 and 5 years
Rate of patients with transient ischemic attack | 1, 2 and 5 years
  Transient ischemic attack at 1, 2 and 5 years
Rate of patients with pulmonary embolism | 1, 2 and 5 years
  Pulmonary embolism at 1, 2 and 5 years
All-cause mortality | 1, 2 and 5 years
  All-cause mortality at 1, 2 and 5 year(s)
LVT size/resolution | 5 years
  LVT size/resolution at follow-up imaging

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Gräni, Prof. PHD, Principal Investigator — Department of Cardiology, University Hospital Bern
Locations (1):
- Department of Cardiology, University Hospital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No